CLINICAL TRIAL: NCT00631059
Title: Assessment and Determination of Chemotherapy Resistance in Newly-Diagnosed or First Relapse Leukemia Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Haluted due to slow accrual
Sponsor: University of California, Irvine (Other)
Responsible Party: Leonard Sender, M.D., Chao Family Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 07-46; HS# 2007-6051
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Leukemia
Keywords: Hitachi; Leukemia; Relapse; Chemotherapy Resistance
MeSH Terms: conditions — Leukemia; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Hem(A)+ Technology — The purpose of the study is to test patients blood. A blood draw will be taken and examined with Hem(A)+ technology.

SUMMARY:
The objective of this protocol is to collect leukemia cell specimens from adults (18 years of age) diagnosed with acute leukemia at time of initial diagnosis and, if applicable, at time of first relapse. These specimens, in conjunction with a de-identified data set, will be utilized prospectively to determine potential chemotherapy resistance in this patient population.

The specific aims of this study are as follows:

To collect peripheral blood specimens from patients diagnosed with acute leukemia at time of initial diagnosis and, if applicable, at time of first relapse To evaluate the leukemia cells in the blood specimens for chemotherapy resistance utilizing the Hem(A)+ technology

To develop a body of evidence from acute leukemia patients that demonstrates the applicability of the Hem(A)+ assay to determine the following:

Predict responders and non-responders to common chemotherapeutic agents Track treatment results and comparison to prediction results from the assay Identify optimal chemotherapy doses for each patient Identify the most efficacious pharmaceutical agent combinations

ELIGIBILITY:
Inclusion Criteria:

Newly Diagnosed Subjects

* The subject is male or female, aged 18 years of age or older
* The subject has a diagnosis of acute lymphocytic leukemia (ALL) or acute myelogenous leukemia (AML); the subject must have a pathology-confirmed diagnosis
* The subject must have a pathology-confirmed diagnosis
* Acute lymphocytic leukemia (ALL) or acute myelogenous leukemia (AML) is defined as having >25% blasts in the bone marrow and/or peripheral blood
* The subject has not received any chemotherapy or treatment for their acute leukemia prior to the initial study visit
* The subject is able and willing to provide written informed consent
* The subject is able to understand the study and cooperate with all study instructions

Relapsed Subjects

* The subject is male or female, aged 18 years of age or older
* The subject has a diagnosis of relapsed acute lymphocytic leukemia (ALL) or relapsed acute myelogenous leukemia (AML)
* The subject must have a pathology-confirmed diagnosis
* Acute lymphocytic leukemia (ALL) or acute myelogenous leukemia (AML) is defined as having ≥ 25% blasts in the bone marrow and/or peripheral blood
* The subject has received one or more of the pre-identified chemotherapeutic agents for treatment of their initial acute leukemia diagnosis
* The subject has not received any systemic chemotherapy or treatment for their relapsed acute leukemia
* Receipt of intrathecal chemotherapy will be permissible
* The subject is able and willing to provide written informed consent
* The subject is able to understand the study and cooperate with all study instructions

Exclusion Criteria:

* The subject has an uncontrolled serious medical or psychiatric illness that, in the opinion of the investigator, would compromise the subject's safety or collection of data
* The subject received treatment with an investigational drug within two weeks of the initial or subsequent study visits
* Subjects under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To collect peripheral blood specimens from patients diagnosed with acute leukemia at time of initial diagnosis and, if applicable, at time of first relapse | No Projected Closing Date

SECONDARY OUTCOMES:
To evaluate the leukemia cells in the blood specimens for chemotherapy resistance utilizing the Hem(A)+ technology | No Projected Closing Date
To develop a body of evidence from acute leukemia patients that demonstrates the applicability of the Hem(A)+ assay | No Projected Closing Date

CONTACTS AND LOCATIONS:
Overall Officials: Leonard S. Sender, MD, Principal Investigator — UCI Department of Medicine -- Hematology/Oncology
Locations (1):
- University of California, Irvine, Orange, California, United States